CLINICAL TRIAL: NCT04734587
Title: Assessment of Silent Brain Injury in Chronic Total Occlusion Patients With Percutaneous Coronary Intervention
Brief Title: Evaluation of Brain Damage Due to Coronary Angioplasty in Percutaneous Intervention Patients
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Muhammet Uyanik, Principal Investigator, Ondokuz Mayıs University
Other Study IDs: SBI IN CTO INTERVENTION
Record Dates: First submitted 2021-01-23; First posted 2021-02-02 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Silent Stroke; Coronary Disease
Keywords: silent brain injury; chronic total occlusion; percutaneous coronary intervention; Neuron specific enolase
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Total Occlusion: Chronic total occlusion patients undergoing percutaneous coronary intervention.
  Interventions: Diagnostic Test: Blood serum Neuron-specific Enolase measurement
- Non-Chronic Total Occlusion: Non-Chronic total occlusion patients undergoing percutaneous coronary intervention.
  Interventions: Diagnostic Test: Blood serum Neuron-specific Enolase measurement

INTERVENTIONS:
Diagnostic Test: Blood serum Neuron-specific Enolase measurement — The Silent Brain Injury ratio was compared by measuring the Neuron-specific enzyme level with venous blood sampling from both patient groups before and after percutaneous coronary intervention.

SUMMARY:
This study examines the formation mechanism and patient-related factors of silent cerebral infarcts, whose importance has become increasingly recognized in patients undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
This study was produced from the assistant's thesis and was previously accepted as a poster at EuroPCR 2020. We recently completed the full-length article.

This thesis study was supported by Ondokuzmayis University.

ELIGIBILITY:
Inclusion Criteria:

* CTO and Non-CTO patients undergoing percutaneous coronary intervention

Exclusion Criteria:

* baseline NSE elevation
* acute coronary syndromes or cardiac surgery within 4 weeks
* patients with a cerebrovascular accident
* intracranial hemorrhage
* and head trauma
* central nervous system tumor
* degenerative central nervous system disorders and neuroendocrine tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were planned to have revascularization due to CTO in at least one coronary artery (CTO Group) and patients who were scheduled for single-vessel elective coronary intervention other than CTO were defined as Non-CTO (control group).
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Baseline Neuron-specific Enolase (NSE) measurement | NSE blood levels were measured 1-2 hours before the procedure.
  Baseline NSE measurement to exclude non-PCI dependent brain injury. Elevation of >20 ng/ml was considered as silent brain injury. Patients with basal nse elevation were considered as SBI and excluded from the study.
Silent Brain Injury diagnosis | 12-18 hours after percutaneous coronary intervention
  NSE blood levels were measured 12-18 hours after the procedure. Elevation of >20 ng/ml was considered as SBI.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Uyanık, M.D., Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuzmayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided